CLINICAL TRIAL: NCT07027280
Title: Noninvasive Intratumor Heterogeneity Evaluation in HNSCC With Multi-omics Insights and Therapeutic Targets
Brief Title: Noninvasive Intratumor Heterogeneity Evaluation in HNSCC
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, xinwei Chen, PHD, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: xChen
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training set
- Test set
- Pathological set

SUMMARY:
This study focuses on tumor heterogeneity, a core challenge in the field of oncology, and innovatively utilizes patient imaging data to deeply mine and analyze intratumoral heterogeneity. By constructing an imaging analysis model for tumor heterogeneity and associating this model with clinical, pathological, transcriptomic, and metabolomic data of patients, a multi-omics decoding of tumor heterogeneity is achieved. The main questions it aims to address are:

Can the ITH model stratify patients' treatment efficacy and prognosis assessment? Can pathological and multi-omics sequencing map the mechanisms behind the ITH model?

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed head and neck squamous cell carcinoma (HNSCC). Complete clinical, imaging, and pathological data. Available complete follow-up information.

Exclusion Criteria:

Patients who received chemotherapy or radiotherapy before surgery. Poor image quality. Tumors too small to be easily identified. History of other concurrent malignant tumors.

Ages: 15 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed HNSCC were collected from the Department of Otolaryngology, the First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
AUC | through study completion, an average of 1 year
C-index | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to the high emphasis on patient privacy protection, there is currently no information about public availability of the dataset in this study. After the relevant articles of this study are officially published, peers can apply to obtain the research data from the corresponding author for legitimate scientific research purposes.